CLINICAL TRIAL: NCT03173703
Title: Random, Controlled, Single-blinded, Multi-center and Non-inferiority Clinical Study to Evaluate Safety and Effectiveness of XenoSure® Biological Patch in the Application of Peripheral Vascular Repair
Brief Title: Evaluate Safety and Effectiveness of XenoSure® Biological Patch in the Application of Peripheral Vascular Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LeMaitre Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P15077-2
Record Dates: First submitted 2017-05-25; First posted 2017-06-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Arm (Experimental): Test Arm are subjects to be implanted with test article -XenoSure patch. The interventions include: Repair/reconstruction of the diseased vessel; Implant the XenoSure patch
  Interventions: Device: Implant the XenoSure patch; Procedure: Repair/reconstruction of the diseased vessel
- Control Arm (Active Comparator): Test Arm are subjects to be implanted with B. Braun's Vascular-Patch.The interventions include: Repair/reconstruction of the diseased vessel; Implant the Vascular-Patch.
  Interventions: Procedure: Repair/reconstruction of the diseased vessel; Device: Implant the Vascular-Patch

INTERVENTIONS:
Device: Implant the XenoSure patch — The LeMaitre XenoSure patch will be used when close the repaired vessel
  Arms: Test Arm
Procedure: Repair/reconstruction of the diseased vessel — The diseased vessel is surgically repaired such as removing the clots.
Device: Implant the Vascular-Patch — The B. Braun Vascular-Patch will be used when close the repaired vessel
  Arms: Control Arm

SUMMARY:
The purpose of this trial is to collect safety and effectiveness data to support peripheral vascular indication of XenoSure biologic patch. This trial is performed to meet the China FDA regulation in this kind of device. The clinical trial will be performed solely inside China under GCP regulation and all applicable China regulations on medical device clinical trial.

DETAILED DESCRIPTION:
The purpose of this trial is to collect safety and effectiveness data to support peripheral vascular indication of XenoSure biologic patch. This trial is performed to meet the China FDA regulation in this kind of device. The clinical trial will be performed solely inside China under GCP regulation and all applicable China regulations on medical device clinical trial.

144 subjects for peripheral vascular repair, including respective 72 subjects for the trial group and the control group.

ELIGIBILITY:
Inclusion Criteria:

- 1) Any man or woman aged between 18~80 years old 2) The expected lifetime of no less than 12 months 3) The subject can be considered for suturing with XenoSure Biological Patch after the peripheral vascular repair surgery. The subject's targeted arterial diameter is less than 5mm or the arterial incision length is more than 4cm and less than 9cm.

4) Physical conditions and vital signs meet requirements for the surgery. 5) The subjects and/or their guardians sign the written Informed Consent Form.

Exclusion Criteria:

1. Patients with severe visceral diseases in heart, liver, kidney, etc.
2. Patients have unstable vital signs and not suitable for the surgery indications
3. Patients need vascular outflow stenting repair in the same location with XenoSure® Biological Patch.
4. Pregnant or lactating women
5. Patients With severe allergic history (especially allergic to bovine materials)
6. Patients with the past medical history of severe immunodeficiency disease
7. The subject has used or plans to use immunomodulatory drugs for more than half a year.
8. The subject with poor blood clotting function is defined as that pre-operative INR or APTT is prolonged over 30% than the reference value without drug intervention, or that blood platelet count is less than 100*10^9/L.
9. The subject has severe kidney disorders or diseases with the estimated glomerular filtration rate [GRF]<30mL/min/1.73m2.
10. The subject's ALT or AST level is 2.5 times higher than the upper normal limit or the subject has active liver disease or icterus.
11. The subject has participated in another clinical study within 3 months or is participating in another clinical study now.
12. The investigator believes that the subject has other reasons unsuitable for inclusion.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Primary patency measured by ultrasound | 6 months
  The treated vessel is considered "patent" if the re-narrowing of the ID of the vessel is less than 20% of the ID that measured immediately after procedure. The study is considered achieved its primary endpoint if the primary patency rate of test device is non-inferior to the rate of the comparator device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hua Shan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No